CLINICAL TRIAL: NCT05800925
Title: Triage Survey for Psychiatry Research Eligibility
Acronym: TRIAGE-Psych
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adams Clinical (Network)
Responsible Party: Sponsor
Other Study IDs: TRIAGE-Psych-101
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder; Borderline Personality Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Borderline Personality Disorder; Generalized Anxiety Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Participants will be surveyed on demographics, medical history, and current psychiatric symptoms. Vital signs, urine drug screens, and urine pregnancy tests may be collected.

SUMMARY:
TRIAGE-Psych is a survey study designed to assess potential participants' eligibility to screen for industry-sponsored psychiatry clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Participant or Legally Authorized Representative has signed an ICF prior to study-specific procedures being performed.
* Participant is at least 18 years old.

Exclusion Criteria:

* Participant is pregnant, breast-feeding, or planning to become pregnant.
* History of a clinically significant illness which in the investigator's opinion may impact participant safety or the ability to analyze study results.
* Participant represents an acute suicidal risk, as defined as a "yes" response to ideation on C-SSRS questions 4 or 5, or answer "yes" to behavior questions within 90 days of screening.
* Moderate or severe substance use disorder within 90 days prior to screen, according to DSM-5 criteria that in the investigator's opinion could pose undue risk to the participant.
* Any condition that in the investigator's opinion makes a participant unsuitable for the study.
* Currently employed by Adams Clinical or a first-degree relative of an employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of any sex, age 18+, who have expressed interest in participating in an industry-sponsored clinical trial of an investigational product for indications in psychiatry will be screened for clinical appropriateness for a study trial.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who are eligible for industry-sponsored clinical trials, as defined as those who go on to screen for a study | Up to 52 weeks

SECONDARY OUTCOMES:
The proportion of participants who enroll in industry-sponsored clinical trials | Up to 52 weeks
The prevalence of disqualifying comorbid conditions that prevent screening or enrollment in industry-sponsored clinical trials | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Copley Clinical, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Berman Clinical, New York, New York